CLINICAL TRIAL: NCT00089011
Title: A Multi-Center Study of Nonmyeloablative Conditioning With TBI or Fludarabine/TBI for HLA-matched Related Hematopoietic Cell Transplantation for Treatment of Hematologic Malignancies With Post Grafting Immunosuppression With Tacrolimus and Mycophenolate Mofetil
Brief Title: Tacrolimus and Mycophenolate Mofetil in Preventing Graft-Versus-Host Disease in Patients Who Have Undergone Total-Body Irradiation With or Without Fludarabine Phosphate Followed by Donor Peripheral Blood Stem Cell Transplant for Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1898.00; NCI-2010-00267 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1898.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P01CA078902 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Results first posted 2017-05-22 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2019-12

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Blastic Phase Chronic Myelogenous Leukemia; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Burkitt Lymphoma; Childhood Chronic Myelogenous Leukemia; Childhood Diffuse Large Cell Lymphoma; Childhood Immunoblastic Large Cell Lymphoma; Childhood Myelodysplastic Syndromes; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Chronic Phase Chronic Myelogenous Leukemia; Contiguous Stage II Adult Burkitt Lymphoma; Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Contiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Contiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Contiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Contiguous Stage II Adult Lymphoblastic Lymphoma; Contiguous Stage II Grade 1 Follicular Lymphoma; Contiguous Stage II Grade 2 Follicular Lymphoma; Contiguous Stage II Grade 3 Follicular Lymphoma; Contiguous Stage II Mantle Cell Lymphoma; Contiguous Stage II Marginal Zone Lymphoma; Contiguous Stage II Small Lymphocytic Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; de Novo Myelodysplastic Syndromes; Essential Thrombocythemia; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Polycythemia Vera; Post-transplant Lymphoproliferative Disorder; Previously Treated Myelodysplastic Syndromes; Primary Myelofibrosis; Prolymphocytic Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Refractory Multiple Myeloma; Relapsing Chronic Myelogenous Leukemia; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage I Adult Burkitt Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Stage I Adult Diffuse Mixed Cell Lymphoma; Stage I Adult Diffuse Small Cleaved Cell Lymphoma; Stage I Adult Immunoblastic Large Cell Lymphoma; Stage I Adult Lymphoblastic Lymphoma; Stage I Adult T-cell Leukemia/Lymphoma; Stage I Childhood Anaplastic Large Cell Lymphoma; Stage I Childhood Large Cell Lymphoma; Stage I Childhood Lymphoblastic Lymphoma; Stage I Childhood Small Noncleaved Cell Lymphoma; Stage I Chronic Lymphocytic Leukemia; Stage I Cutaneous T-cell Non-Hodgkin Lymphoma; Stage I Grade 1 Follicular Lymphoma; Stage I Grade 2 Follicular Lymphoma; Stage I Grade 3 Follicular Lymphoma; Stage I Mantle Cell Lymphoma; Stage I Marginal Zone Lymphoma; Stage I Multiple Myeloma; Stage I Small Lymphocytic Lymphoma; Stage IA Mycosis Fungoides/Sezary Syndrome; Stage IB Mycosis Fungoides/Sezary Syndrome; Stage II Adult T-cell Leukemia/Lymphoma; Stage II Childhood Anaplastic Large Cell Lymphoma; Stage II Childhood Large Cell Lymphoma; Stage II Childhood Lymphoblastic Lymphoma; Stage II Childhood Small Noncleaved Cell Lymphoma; Stage II Chronic Lymphocytic Leukemia; Stage II Cutaneous T-cell Non-Hodgkin Lymphoma; Stage II Multiple Myeloma; Stage IIA Mycosis Fungoides/Sezary Syndrome; Stage IIB Mycosis Fungoides/Sezary Syndrome; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Adult T-cell Leukemia/Lymphoma; Stage III Childhood Anaplastic Large Cell Lymphoma; Stage III Childhood Large Cell Lymphoma; Stage III Childhood Lymphoblastic Lymphoma; Stage III Childhood Small Noncleaved Cell Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Multiple Myeloma; Stage III Small Lymphocytic Lymphoma; Stage IIIA Mycosis Fungoides/Sezary Syndrome; Stage IIIB Mycosis Fungoides/Sezary Syndrome; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Childhood Anaplastic Large Cell Lymphoma; Stage IV Childhood Large Cell Lymphoma; Stage IV Childhood Lymphoblastic Lymphoma; Stage IV Childhood Small Noncleaved Cell Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma; Stage IVA Mycosis Fungoides/Sezary Syndrome; Stage IVB Mycosis Fungoides/Sezary Syndrome; Testicular Lymphoma; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Adult Acute Myeloid Leukemia; Untreated Childhood Acute Lymphoblastic Leukemia; Untreated Childhood Acute Myeloid Leukemia and Other Myeloid Malignancies; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Blast Crisis; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Leukemia, Myeloid, Chronic-Phase; Thrombocythemia, Essential; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Polycythemia Vera; Primary Myelofibrosis; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Leukemia, Hairy Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — fludarabine phosphate; Whole-Body Irradiation; Mycophenolic Acid; Tacrolimus; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (nonmyeloablative conditioning with fludarabine and TBI) (Experimental): Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  Interventions: Drug: fludarabine phosphate; Radiation: total-body irradiation; Other: laboratory biomarker analysis
- Arm II (nonmyeloablative conditioning with TBI) (Experimental): Patients undergo TBI on day 0. All patients then undergo allogeneic peripheral blood stem cell transplantation on day 0 and receive tacrolimus PO every 12 hours on days -3 to 180, with taper on day 56, or tacrolimus IV if unable to tolerate PO; and mycophenolate mofetil PO every 12 hours on days 0-27 or mycophenolate mofetil IV if unable to tolerate PO.
  Interventions: Radiation: total-body irradiation; Drug: mycophenolate mofetil; Drug: tacrolimus; Procedure: peripheral blood stem cell transplantation; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
  Arms: Arm I (nonmyeloablative conditioning with fludarabine and TBI)
Radiation: total-body irradiation — Undergo radiotherapy
  Other Names: TBI
Drug: mycophenolate mofetil — Given IV or PO
  Other Names: Cellcept; MMF
  Arms: Arm II (nonmyeloablative conditioning with TBI)
Drug: tacrolimus — Given IV or PO
  Other Names: FK 506; Prograf
  Arms: Arm II (nonmyeloablative conditioning with TBI)
Procedure: peripheral blood stem cell transplantation — Undergo allogeneic peripheral blood stem cell transplant
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
  Arms: Arm II (nonmyeloablative conditioning with TBI)
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation — Undergo allogeneic peripheral blood stem cell transplant
  Arms: Arm II (nonmyeloablative conditioning with TBI)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well tacrolimus and mycophenolate mofetil works in preventing graft-versus-host disease in patients who have undergone total-body irradiation (TBI) with or without fludarabine phosphate followed by donor peripheral blood stem cell transplant for hematologic cancer. Giving low doses of chemotherapy, such as fludarabine phosphate, and TBI before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving tacrolimus and mycophenolate mofetil after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the incidence of grade III/IV graft-versus-host disease (GVHD) after conditioning with 200 centigray (cGy) TBI alone or Fludarabine (fludarabine phosphate)/200 cGy TBI followed by tacrolimus (Tac)/mycophenolate mofetil (MMF) immunosuppression in patients with hematologic malignancies.

II. To estimate the incidence of chronic extensive GVHD.

SECONDARY OBJECTIVES:

I. To estimate the incidences of graft rejection.

II. To estimate overall survival 1-year after conditioning.

III. To evaluate the incidences of grades II-IV acute GVHD.

IV. To evaluate the rates of disease progression and/or relapse-related mortality.

V. To estimate the rate and duration of steroid use for the treatment of chronic GVHD.

OUTLINE: Patients are assigned to 1 of 2 treatment arms.

ARM I (nonmyeloablative conditioning with fludarabine phosphate and TBI): Patients receive fludarabine phosphate intravenously (IV) on days -4 to -2 and undergo TBI on day 0.

ARM II (nonmyeloablative conditioning with TBI): Patients undergo TBI on day 0.

All patients then undergo allogeneic peripheral blood stem cell transplantation on day 0 and receive tacrolimus orally (PO) every 12 hours on days -3 to 180, with taper on day 56, or tacrolimus IV if unable to tolerate PO; and mycophenolate mofetil PO every 12 hours on days 0-27 or mycophenolate mofetil IV if unable to tolerate PO.

Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 2 years and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be not eligible for conventional allogeneic hematopoietic cell transplantation (HCT) and must have disease expected to be stable for at least 100 days without chemotherapy; patients with hematologic malignancies treatable with HCT or with a B cell malignancy except those curable with autologous transplant will be included; patients not eligible for active disease specific protocols may be enrolled in this protocol; patients will include the following
* Diffuse large B cell non-Hodgkin lymphoma (NHL) and other aggressive lymphomas - not eligible for conventional myeloablative HCT or after autologous HCT
* Low grade NHL- with < 6 months duration of complete response (CR) between courses of conventional therapy
* Mantle cell NHL- may be treated in first CR
* Chronic lymphocytic leukemia (CLL) - must have either 1) failed to meet National Cancer Institute (NCI) Working Group criteria for complete or partial response after therapy with a regimen containing fludarabine phosphate (FLU) (or another nucleoside analog, e.g. 2-chlorodeoxyadenosine [2-CDA], pentostatin) or experience disease relapse within 12 months after completing therapy with a regimen containing FLU (or another nucleoside analog); 2) failed FLU-cyclophosphamide (CY)-Rituximab (FCR) combination chemotherapy at any time point; or 3) have "17p deletion" cytogenetic abnormality; patients should have received induction chemotherapy but could be transplanted in 1st CR; 4) patients with a diagnosis of CLL (or small lymphocytic lymphoma) or a diagnosis of CLL that progresses to prolymphocytic leukemia (PLL), or T-cell CLL or PLL
* Hodgkin lymphoma (HL) - must have received and failed frontline therapy; patients must have failed or were not eligible for autologous transplant
* Multiple myeloma (MM) - following a planned autologous transplant or equivalent high-dose therapy without a graft, or following a failed prior autograft
* Acute myeloid leukemia (AML) - must have < 5% marrow blasts at the time of transplant
* Acute lymphoblastic leukemia (ALL) - must have < 5% marrow blasts at the time of transplant
* Chronic myelogenous leukemia (CML) - patients will be accepted beyond first chronic phase (CP1) if they have received previous myelosuppressive chemotherapy or HCT, and have < 5% marrow blasts at time of transplant
* Myelodysplastic syndromes/myeloproliferative disorders (MDS/MPD) - must have received previous myelosuppressive chemotherapy or HCT, and have < 5% marrow blasts at time of transplant
* Waldenstrom's macroglobulinemia - must have failed 2 courses of therapy
* Myelosuppressive chemotherapy must be discontinued three weeks prior to conditioning with the exception of hydroxyurea or imatinib
* Patients < 12 years old must be approved by both the participating institutions' patient review committee such as the Patient Care Conference (PCC) at the Fred Hutchinson Cancer Research Center (FHCRC) and the FHCRC principal investigator
* Patient who refused to be treated on a conventional HCT protocol; for this inclusion criterion, transplants must be approved by both the participating institution's patient review committee such as the Patient Care Conference (PCC) at the FHCRC and the FHCRC principal investigators
* Patients with human leukocyte antigen (HLA)-matched related donors
* Patients with renal failure are eligible; however, patients with renal compromise (serum creatinine > 2.0) will likely have further compromise in renal function and may require hemodialysis (which may be permanent) due to the need to maintain adequate serum tacrolimus levels
* DONOR: Related donor who is HLA genotypically identical at least at one haplotype and may be phenotypically or genotypically identical at the allele level at HLA-A, -B, -C, -DRB1, and -DQB1
* DONOR: Donor must consent to filgrastim (G-CSF) administration and leukapheresis
* DONOR: Donor must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral, subclavian)

Exclusion Criteria:

* Eligible for a high priority curative autologous transplant
* Patient with rapidly progressive, aggressive NHL unless in minimal disease state
* Patients with chronic myelomonocytic leukemia (CMML)
* Life expectancy severely limited by diseases other than malignancy
* Any current central nervous system (CNS) involvement with disease refractory to intrathecal chemotherapy
* Presence of circulating leukemic blasts (in the peripheral blood) detected by standard pathology for patients with AML, ALL or CML
* Fertile men or women unwilling to use contraceptives during and for up to 12 months post treatment
* Female patients who are pregnant or breastfeeding
* Human immunodeficiency virus (HIV)-positive patients
* Patients with active non-hematologic malignancies (except non-melanoma skin cancers); this exclusion does not apply to patients with non-hematologic malignancies that do not require therapy
* Patients with a history of non-hematologic malignancies (except non-melanoma skin cancers) currently in a complete remission, who are less than 5 years from the time of complete remission, and have a > 20% risk of disease recurrence; this exclusion does not apply to patients with non-hematologic malignancies that do not require therapy
* Fungal pneumonia with radiological progression after receipt of amphotericin formulation or mold-active azoles for greater than 1 month
* Karnofsky score < 50 for adult patients
* Lansky-Play performance score < 50 for pediatric patients
* Symptomatic coronary artery disease or ejection fraction < 35% or other cardiac failure requiring therapy (or, if unable to obtain ejection fraction, shortening fraction of < 26%); ejection fraction is required if age > 50 years or there is a history of anthracycline exposure or history of cardiac disease; patients with a shortening fraction < 26% may be enrolled if approved by a cardiologist
* Poorly controlled hypertension
* Diffusing capacity of the lung for carbon monoxide (DLCO) < 30%, total lung capacity (TLC) < 30%, forced expiratory volume in one second (FEV1) < 30% and/or receiving supplementary continuous oxygen; the FHCRC principal investigator (PI) of the study must approve enrollment of all patients with pulmonary nodules
* Liver function abnormalities: Patients with clinical or laboratory evidence of liver disease would be evaluated for the cause of liver disease, its clinical severity in terms of liver function, and the degree of portal hypertension; patients will be excluded if they are found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension or bridging fibrosis, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, and symptomatic biliary disease
* Patients with active bacterial or fungal infections unresponsive to medical therapy
* DONOR: Age less than 12 years
* DONOR: Identical twin
* DONOR: Pregnancy
* DONOR: Infection with HIV
* DONOR: Known allergy to filgrastim (G-CSF)
* DONOR: Current serious systemic illness that would result in increased risk for G-CSF mobilization and harvest of peripheral blood stem cells (PBSC)

Max Age: 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2004-04 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Maloney, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (5):
- United States (4):
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - VA Puget Sound Health Care System, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
- University of Torino, Torino, Italy

REFERENCES:
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Nonmyeloablative Conditioning With Fludarabine and TBI) | Arm II (Nonmyeloablative Conditioning With TBI)
Started | 100 | 50
Completed | 100 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Nonmyeloablative Conditioning With Fludarabine and TBI) | Arm II (Nonmyeloablative Conditioning With TBI) | Total
Number analyzed (Participants) | 100 | 50 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 74 | 49 | 123
  >=65 years | 26 | 1 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 17 | 63
  Male | 54 | 33 | 87
Region of Enrollment [Number; unit: participants]
  United States | 98 | 46 | 144
  Italy | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Grade III/IV GVHD
Description: Number of patients who developed acute/chronic GVHD post-transplant. aGVHD Stages
  Skin:
  a maculopapular eruption involving < 25% BSA a maculopapular eruption involving 25 - 50% BSA generalized erythroderma generalized erythroderma with bullous formation and often with desquamation
  Liver:
  bilirubin 2.0 - 3.0 mg/100 mL bilirubin 3 - 5.9 mg/100 mL bilirubin 6 - 14.9 mg/100 mL bilirubin > 15 mg/100 mL
  Gut:
  Diarrhea is graded 1 - 4 in severity. Nausea and vomiting and/or anorexia caused by GVHD is assigned as 1 in severity. The severity of gut involvement is assigned to the most severe involvement noted. Patients with visible bloody diarrhea are at least stage 2 gut and grade 3 overall.
  aGVHD Grades Grade III: Stage 2 - 4 gut involvement and/or stage 2 - 4 liver involvement Grade IV: Pattern and severity of GVHD similar to grade 3 with extreme constitutional symptoms or death
Time Frame: Day 180 post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nonmyeloablative Conditioning With Fludarabine and TBI) | Arm II (Nonmyeloablative Conditioning With TBI)
Number analyzed (Participants) | 100 | 50
Participants | 2 | 4

2. Primary Outcome: Incidence of Chronic Extensive GVHD
Description: Number of patients who developed chronic extensive GVHD post-transplant. The diagnosis of chronic GVHD requires at least one manifestation that is distinctive for chronic GVHD as opposed to acute GVHD. In all cases, infection and others causes must be ruled out in the differential diagnosis of chronic GVHD.
Time Frame: Day 180 post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nonmyeloablative Conditioning With Fludarabine and TBI) | Arm II (Nonmyeloablative Conditioning With TBI)
Number analyzed (Participants) | 100 | 50
Participants | 15 | 6

3. Secondary Outcome: Incidences of Graft Rejection
Description: Number of patients who rejected their graft. Rejection is defined as the inability to detect or loss of detection of greater than 5% donor T cells (CD3+) as a proportion of the total T cell population, respectively, after nonmyeloablative HCT.
Time Frame: Day 180 post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nonmyeloablative Conditioning With Fludarabine and TBI) | Arm II (Nonmyeloablative Conditioning With TBI)
Number analyzed (Participants) | 100 | 50
Participants | 0 | 0

4. Secondary Outcome: Overall Survival
Description: Number of patients surviving post-transplant.
Time Frame: At 1 year after conditioning
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nonmyeloablative Conditioning With Fludarabine and TBI) | Arm II (Nonmyeloablative Conditioning With TBI)
Number analyzed (Participants) | 100 | 50
Participants | 85 | 39

5. Secondary Outcome: Incidences of Grades II-IV Acute GVHD
Description: Number of patients who developed acute/chronic GVHD post-transplant. aGVHD Stages
  Skin:
  a maculopapular eruption involving < 25% BSA a maculopapular eruption involving 25 - 50% BSA generalized erythroderma generalized erythroderma with bullous formation and often with desquamation
  Liver:
  bilirubin 2.0 - 3.0 mg/100 mL bilirubin 3 - 5.9 mg/100 mL bilirubin 6 - 14.9 mg/100 mL bilirubin > 15 mg/100 mL
  Gut:
  Diarrhea is graded 1 - 4 in severity. Nausea and vomiting and/or anorexia caused by GVHD is assigned as 1 in severity. The severity of gut involvement is assigned to the most severe involvement noted. Patients with visible bloody diarrhea are at least stage 2 gut and grade 3 overall.
  aGVHD Grades Grade II: Stage 1 - 3 skin and/or stage 1 gut involvement and/or stage 1 liver involvement Grade III: Stage 2 - 4 gut involvement and/or stage 2 - 4 liver involvement Grade IV: Pattern and severity of GVHD similar to grade 3 with extreme constitutional symptoms or death
Time Frame: Day 180 post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nonmyeloablative Conditioning With Fludarabine and TBI) | Arm II (Nonmyeloablative Conditioning With TBI)
Number analyzed (Participants) | 100 | 50
Participants | 26 | 14

6. Secondary Outcome: Rates of Disease Progression
Description: Relapse/Progression criteria:
  CML New cytogenetic abnormality and/or development of accelerated phase or blast crisis. The criteria for accelerated phase will be defined as unexplained fever >38.3°C, new clonal cytogenetic abnormalities in addition to a single Ph-positive chromosome, marrow blasts and promyelocytes >20%.
  CMML, AML, ALL >30% BM blasts w/ deteriorating performance status, or worsening of anemia, neutropenia, or thrombocytopenia.
  CLL ≥1 of: Physical exam/imaging studies ≥50% increase or new, circulating lymphocytes by morphology and/or flow cytometry ≥50% increase, and lymph node biopsy w/ Richter's transformation.
  NHL >25% increase in the sum of the products of the perpendicular diameters of marker lesions, or the appearance of new lesions.
  MM
  ≥100% increase of the serum myeloma protein from its lowest level, or reappearance of myeloma peaks that had disappeared w/ treatment; or definite increase in the size or number of plasmacytomas or lytic bone lesions.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nonmyeloablative Conditioning With Fludarabine and TBI) | Arm II (Nonmyeloablative Conditioning With TBI)
Number analyzed (Participants) | 100 | 50
Participants | 41 | 33

7. Secondary Outcome: Rates of Relapse-related Mortality
Description: Number of patients who expired with relapsed/progressive disease.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nonmyeloablative Conditioning With Fludarabine and TBI) | Arm II (Nonmyeloablative Conditioning With TBI)
Number analyzed (Participants) | 100 | 50
Participants | 28 | 23

8. Secondary Outcome: Rate and Duration of Steroid Use for the Treatment of Chronic GVHD
Description: Number of patients that received prednisone treatment of chronic GVHD, and number of days for which they received prednisone.
Time Frame: Up to 5 years
Population: Only those patients who received steroids for treatment of chronic GVHD.
Measure: Median (Full Range); unit: days
Arm/Group | Arm I (Nonmyeloablative Conditioning With Fludarabine and TBI) | Arm II (Nonmyeloablative Conditioning With TBI)
Number analyzed (Participants) | 44 | 21
days | 78 [1 to 1156] | 89 [1 to 420]

ADVERSE EVENTS:
Arm/Group | Arm I (Nonmyeloablative Conditioning With Fludarabine and TBI) | Arm II (Nonmyeloablative Conditioning With TBI)
Serious Adverse Events (participants affected / at risk) | 8/100 | 5/50
Other Adverse Events (participants affected / at risk) | 28/100 | 17/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Nonmyeloablative Conditioning With Fludarabine and TBI) (N=100) | Arm II (Nonmyeloablative Conditioning With TBI) (N=50)
Death, Renal Failure, Cardiac Failure (Cardiac disorders) | 1 | 0
Death due to severe refractory autoimmune hemolytic anemia (present prior to transplant) (Immune system disorders) | 1 | 0
Death, elevated bilirubin, fevers (Hepatobiliary disorders) | 1 | 0
Right central artery occlusion with right eye blindness (Eye disorders) | 1 | 0
Severe abdominal pain due to gut GVHD and supravantricular arrhythmia/Atrial fibrillation (Immune system disorders) | 1 | 0
Mental Status Change while on ativan, oxycodone, and flexeril (Psychiatric disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Elevated LFT's with rising total bilirubin level (Hepatobiliary disorders) | 1 | 0
Hypoxia and Hypotension (Vascular disorders) | 0 | 1
Death, secondary to sepsis with multiorgan failure (Infections and infestations) | 0 | 1
Perforated gastric ulcer (Gastrointestinal disorders) | 0 | 1
Death due to adenovirus nephritis, sepsis, multifactorial renal failure (Infections and infestations) | 0 | 1
Elevated creatinine level (Renal and urinary disorders) | 0 | 1 — Elevated creatinine level r/t acute renal failure in the setting of chronic kidney disease due to multiple myeloma
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Nonmyeloablative Conditioning With Fludarabine and TBI) (N=100) | Arm II (Nonmyeloablative Conditioning With TBI) (N=50)
Increased Creatinine (Renal and urinary disorders) | 20 | 15
Hemolysis / Hemolytic Anemia (Blood and lymphatic system disorders) | 5 | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 8 | 3
Hypoxia / Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Hypotension (Cardiac disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes